CLINICAL TRIAL: NCT03660111
Title: Establishment of Spirometric Predicted Values in Bolivia
Brief Title: Spirometric Predicted Values in Bolivia
Acronym: SPIROBOLIVIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Giuseppe Liistro, Head of clinics, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPIROBOLIVIA
Record Dates: First submitted 2018-07-03; First posted 2018-09-06 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Spirometry; Respiratory Function Tests
MeSH Terms: interventions — Spirometry

STUDY DESIGN:
Masking Description: subjects will be assigned to their inclusion number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- spirometry (Other): single spirometry: only a routine diagnostic test
  Interventions: Diagnostic Test: spirometry

INTERVENTIONS:
Diagnostic Test: spirometry — only measurement of spirometry

SUMMARY:
There is no local predicted values for spirometry available in Bolivia. The aim of the present study is to establish moderne predicted values for healthy non-smokers recruited in a major city of Bolivia, Santa Cruz De La Sierra.

DETAILED DESCRIPTION:
There is no local predicted values for spirometry available in Bolivia. To establish the predicted spirometric normal values in Bolivia, 500 healthy men and women, non-smokers will be recruited to perfom spirometry using following the actual ATS/ERS 2005 guidelines.

The spirometer is a Bodybox 5500 (Medisoft, Belgium). The tests will be performed by a highly-trained pneumologist, Dr A. Ajata.

Anthropometric variables recorded: age, sex, weight, standing and sitting height.

Spirometric variables recorded: FEV1, FVC, PEF, FEV6, FEF25,50,75 and MEF Statistical anaysis will be done using R and SPSS softwares. Predicted equations will be compared with existing ones, especially the new GLI-2012 predicted equations.

ELIGIBILITY:
Inclusion Criteria:

* healthy and non-smokers

Exclusion Criteria:

* unhealthy smokers
* subjects unable to understand/sign informed consent unable to understand/perform spirometric measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
FEV1 | measurements done one time at recruitment during spirometry
  Forced expiratory volume in one second (Liter)
FVC | measurements done one time at recruitment during spirometry
  forced vital capacity (Liter)
FEV1/FVC ratio | measurements done one time at recruitment during spirometry
  FEV1/FVC ratio , %

SECONDARY OUTCOMES:
Standing height | measurements done one time at recruitment just before spirometry
  Standing height
seated height | measurements done one time at recruitment just before spirometry
  seated height

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica del Pulmón, Santa Cruz, Bolivia

IPD SHARING:
Plan to Share IPD: Yes
All the parts of the study will be available for reviewing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At article submission for reviewing until final acceptation
Access Criteria: Following the reviewers' requirements